CLINICAL TRIAL: NCT07028294
Title: Effectiveness and Clinical Application of Multidisciplinary Combined Exercise and Nutrition Intervention for Sarcopenic Older Adults With Metabolic Syndrome: Multicenter Empirical Study
Brief Title: Multidisciplinary Combined Exercise and Nutrition Intervention for Sarcopenia (2)
Acronym: MENTORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-2010/645-005 (2); RS-2020-KH095863 (Other Grant/Funding Number: Ministry of Health & Welfare, Republic of Korea)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia
Keywords: sarcopenia; older adults; exercise; nutrition; standard intervention
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined exercise and nutrition intervention (Experimental): Customized exercise and nutrition intervention by underlying disease and functional state for 12 weeks during intervention period.
  Interventions: Combination Product: Combined exercise and nutrition intervention

INTERVENTIONS:
Combination Product: Combined exercise and nutrition intervention — Combined exercise and nutrition intervention for 12 weeks (an introductory phase 3 weeks, an expanded phase 3 weeks, and a maintenance phase 6 weeks). Exercise intervention (each 60-min session) includes stretching, resistance exercise, and aerobic exercise according to protocol. Nutritional intervention includes investigating dietary habits and calculate insufficient protein intake using Mini Nutritional Aseessment (MNA) and Korean Protein Assessment Tool (KPAT) to provide customized diet and high protein drink.

SUMMARY:
This is an empirical study, which aims to examine the effect of a 12-week combined exercise-nutrition intervention in older adults with sarcopenia and to provide data for clinical and policy decision-making of sarcopenia. The study conducts the combined exercise-nutrition intervention that was previously carried out as a randomized controlled trial. Hand grip strength, gait speed, knee extensor muscle power, physical performance, muscle mass using DEXA, quality of life, activities of daily living, sarcopenia screening questionnaire, nutritional assessment will be evaluated on baseline, 12-weeks and 24-weeks after intervention.

DETAILED DESCRIPTION:
The definition of sarcopenia is age-related loss of skeletal muscle and physical functions. Sarcopenia is emerging health problem and increases medical expenditure as the population ages. Sarcopenia is closely related to chronic diseases and geriatric diseases. In particular, patients with metabolic syndrome showed a high prevalence of muscle loss and muscle weakness. It has been reported exercise in sarcopenia patients not only improved insulin sensitivity and physical performance but also helped the treatment of the diseases. Also, it has recently demonstrated that combined exercise-nutrition intervention improved muscle function in elderly patients. However, the standard protocol for the combined exercise-nutrition intervention has not been established yet. Therefore, this study aims to see the effects of a 12-week combined exercise-nutrition intervention in sarcopenia patients.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 65 years and under 90 years
* patients who meet the criteria for the Asian Working Group for Sarcopenia (AWGS) 2019
* patients who had metabolic syndrome

Exclusion Criteria:

* patients with less than estimated glomerular filtration rate (eGFR) 30
* patients with musculoskeletal or chronic lung disease incapable of exercise
* patients with untreated or uncontrolled cardiovascular disease which may affect muscle mass or performing exercise
* patients less than 5 years after treatment of malignant tumor
* patients with liver cirrhosis, diabetes and other chronic disease
* patients who cannot perform combined exercise nutrition intervention for other reasons

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
5-times chair stand test | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Change from baseline 5-times chair stand test to 12 weeks after assessment, measured by 5-times chair stand test

SECONDARY OUTCOMES:
Physical performance | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Short Physical Performance Battery [range from 0 to 12 score]
Gait speed test | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  measured by 6 meter gait speed
Appendicular skeletal muscle mass | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  measured using Dual-energy X-ray absorptiometry (DEXA), Bioelectrical impedance analysis (BIA)
Health Related Quality of Life | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of quality of life using EQ-5D [range from 5 to 25 score]. Higher value means worse quality of life
Basic and instrumental activities of daily living | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of basic and instrumental activities of daily living using Korean Activity of Daily Living (K-ADL), Korean Instrumental Activity of Daily Living (K-IADL) [range from 0 to 33]. Low value means poor ability of activities.
Sarcopenia screening questionnaire | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of quality of life using Strength, Assistance with walking, Rising from a chair, Climbing stairs and Falls (SARC-F) questionnair [range from 0 to 10].
Nutritional Assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of nutritional state using Mini-Nutritional Assessment (MNA) [range from 1 to 30 score], Korean Protein Assessment Tool (KPAT)
Handgrip strength | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of hand grip strength using Hand-held dynamometer
Delirium assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of delirium using Delirium Rating Scale (DRS) [range from 0 to 32 score]. Higher value means worse delrious status
Physical acitivity assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Measured by Korean Physical Activity Scale for the Elderly (K-PASE) [range from 0 to 1382.52 score]. Higher value means better physical status
Cognitive assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of cognitive state using Korean Mini Mental Status Examination, 2nd edition (K-MMSE2) [range from 0 to 30 score]
Psychiatric state | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  Evaluation of psychiatric state using Short Form of Geriatric Depression Scale-Korea (SGDS-K) [range from 0 to 30 score]
Swallowing assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  measured by Standardized Swallowing Assessment (SSA)
Empowerment assessment | Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)
  measured by Korean version of Health Empowerment Scale (K-HES) [range from 8 to 40 score]. Higher value means better empowerment status

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Young Lim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nipp RD, Fuchs G, El-Jawahri A, Mario J, Troschel FM, Greer JA, Gallagher ER, Jackson VA, Kambadakone A, Hong TS, Temel JS, Fintelmann FJ. Sarcopenia Is Associated with Quality of Life and Depression in Patients with Advanced Cancer. Oncologist. 2018 Jan;23(1):97-104. doi: 10.1634/theoncologist.2017-0255. Epub 2017 Sep 21. PMID 28935775
- [Background] Malafarina V, Uriz-Otano F, Malafarina C, Martinez JA, Zulet MA. Effectiveness of nutritional supplementation on sarcopenia and recovery in hip fracture patients. A multi-centre randomized trial. Maturitas. 2017 Jul;101:42-50. doi: 10.1016/j.maturitas.2017.04.010. Epub 2017 Apr 22. PMID 28539168
- [Background] Jang HC. How to Diagnose Sarcopenia in Korean Older Adults? Ann Geriatr Med Res. 2018 Jun;22(2):73-79. doi: 10.4235/agmr.2018.22.2.73. Epub 2018 Jun 30. PMID 32743250
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820